CLINICAL TRIAL: NCT01976247
Title: Pilot Study Comparing the Effectiveness of a Noninvasive Cryolipolysis Device vs. a High Intensity Focused Ultrasound Device for Fat Reduction: A Randomized Control Trial
Brief Title: A Pilot Study Testing a Noninvasive Cryolipolysis Device Versus a High Intensity Focused Ultrasound Device for Fat Reduction
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: STU84032
Record Dates: First submitted 2013-10-15; First posted 2013-11-05 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Abdominal Fat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Noninvasive Cryolipolysis Device (Active Comparator): The Zeltiq System is a noninvasive (not breaking the skin) device that reduces fat by freezing fat cells until they break apart.
  Interventions: Device: Noninvasive Cryolipolysis Device
- High Intensity Focused Ultrasound Device (Active Comparator): The LipoSonix System is a noninvasive ultrasound device, which can be used to selectively target and destroy fat tissue located deep under the skin.
  Interventions: Device: High Intensity Focused Ultrasound Device

INTERVENTIONS:
Device: High Intensity Focused Ultrasound Device
  Other Names: Liposonix
  Arms: High Intensity Focused Ultrasound Device
Device: Noninvasive Cryolipolysis Device
  Other Names: Zeltiq
  Arms: Noninvasive Cryolipolysis Device

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of the Zeltiq System and LipoSonix System for fat reduction and improving body shape.

DETAILED DESCRIPTION:
At baseline visit, subjects who meet inclusion and exclusion criteria will be enrolled. Subjects will be randomly assigned to receive Zeltiq treatment to either their right or left flank The contralateral flank will receive Liposonix treatment. A total of three identical treatments will be completed monthly for 3 consecutive months. Subjects will return 4 weeks following the last treatment for follow up photography, measurements, and assessments. This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects ages 30-65 years old.
2. Body mass index (BMI) between 18 and 29.99. (BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches).
3. Subjects are in good health.
4. Willing and able to abstain from partaking in any treatment other than the study procedure (existing or new) to promote body contouring and/or weight loss during the course of study participation.
5. Subjects agree to maintain their weight (i.e. within 5 pounds) by not making any changes to diet or lifestyle during the study.
6. The subjects have the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.

Exclusion Criteria:

1. Pregnant or lactating or intends to become pregnant in the next 9 months.
2. Unable to understand the protocol or to give informed consent.
3. Any previous and/or pending procedures at the treatment area or that may likely affect the treatment area.
4. Pending and/or anticipated major change in diet or exercise pattern in the six weeks following the last treatment or who has taken diet pills within the last 6 months..
5. History of asthma or chronic obstructive pulmonary diseases.
6. Active skin disease or skin infection in the treatment area.
7. Bleeding tendency or coagulopathy.
8. Subjects who are allergic to lidocaine.
9. Any other condition that would, in the professional opinion of the investigator, potentially affect response or participation in the clinical study, or would pose as an unacceptable risk to the subject.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in best overall cosmetic appearance (right side or left side better)rated by a blinded dermatologist from baseline to week 12 | 1 hour at baseline and week 12
  The primary outcome was a blinded rating of the treatment area (Noninvasive Cryolipolysis Device vs. a High Intensity Focused Ultrasound Device) with the best cosmetic appearance. A dermatologist will blindly evaluate the treated areas of each side from live subjects at baseline and on the final follow up visit (week 12).

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States